CLINICAL TRIAL: NCT06147505
Title: Clinical Study of Evaluating the Safety and Initial Efficacy of XS005 Injection Combined With Stupp Regimen for Adjuvant Chemotherapy in Subjects With Primary Glioblastoma(GBM)
Brief Title: XS005 Injection Combined With Stupp Regimen for Adjuvant Chemotherapy in Subjects With Primary Glioblastoma(GBM)
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The hospital is under renovation
Sponsor: Dushu Lake Hospital Affiliated to Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XS-005
Record Dates: First submitted 2023-11-08; First posted 2023-11-27 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2023-11

CONDITIONS: Tumor
Keywords: XS005
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Subjects With Tumor
  Interventions: Biological: XS005 Injection

INTERVENTIONS:
Biological: XS005 Injection — Treatment on this study includes XS005 infusions over an 16 week period. Phase 1： dose escalation (3+3); Phase 2 : dose of recommended phase 2 dose(RP2D).
  Other Names: XS005

SUMMARY:
The main objective of this clinical study is to evaluate the safety of XS005 injection; to determine the maximum tolerated dose . Furthermore, initial efficacy will be examined.

DETAILED DESCRIPTION:
Treatment on this study includes eight XS005 infusions over an 16 week period. The study will evaluate the safety, feasibility and maximum tolerated dose (MTD) of XS005 using a 3+3 study design . The total study duration will be 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years old (including the threshold), both male and female;
2. Expected survival ≥6 months;
3. Karnofsky performance status(KPS) score ≥60 before treatment;
4. The level of organ and bone marrow function must meet the following requirements:

   * Bone marrow: Absolute neutrophil count (ANC) ≥1.5×109/L, platelet count ≥100×109/L, hemoglobin ≥90g/L, and no platelet or red blood cell transfusion within 14 days prior to first administration. And did not receive blood transfusion or biological response regulators (such as granulocyte growth factor, erythrocyte growth factor, interleukin-11, etc.) within 14 days before the first administration;
   * Liver function: No history of cirrhosis (Child-Pugh grade B, C). Serum total bilirubin (TBIL) ≤1.5× upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN;
   * Renal function: serum creatinine ≤1.5×ULN, or creatinine clearance ≥50ml/min (Cockcroft-Gault formula); Qualitative urine protein ≤1+; If the qualitative urine protein is ≥2+, it is necessary to conduct a quantitative urine protein test for 24 hours. According to the examination results, the researchers made the admission judgment.
   * Coagulation function: prothrombin time (PT) ≤1.5×ULN; International standardized ratio (INR) ≤1.5×ULN, and activated partial thromboplastin time (APTT) ≤1.5×ULN (except those receiving therapeutic anticoagulants);
5. The subjects (including male subjects) have no pregnancy plan and voluntarily take effective contraceptive measures during the screening period and from the beginning of the study administration to the last dose of the study drug within 6 months after the study drug is administered, and have no sperm or egg donation plans, in which the study period should voluntarily take effective contraceptive measures;
6. Able to understand the procedures and methods of this study, willing to sign informed consent and strictly follow the clinical study protocol to complete this study.

Exclusion Criteria:

1. Patients who received other anti-tumor drugs (including chemotherapy, targeted drugs other than bevacizumab, immunotherapy, Chinese medicine anti-tumor therapy, etc.) except for patients who received concurrent radiotherapy and chemotherapy for GBM after surgery (TMZ dosage ≤75mg/m2, radiotherapy dose limited to 50-60Gy);
2. Previous or current malignant tumors of other types, except for the following cases: basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin or cervical cancer in situ;
3. The presence of any contraindications to MRI, such as: use of a pacemaker, infusion pump, or allergy to MRI contrast agents;
4. Receive live attenuated vaccine or vaccine within 4 weeks prior to the first study drug treatment or plan to receive live vaccine during the study period;
5. Subjects with active or pre-existing autoimmune diseases that are likely to recur, or patients at high risk (such as those who have received an organ transplant and require immunosuppressive therapy).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-29 (Actual); Primary Completion 2025-11-02 (Estimated); Study Completion 2025-12-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicities (DLTs) | within 7 days after the the first infusion of XS005.
  DLT is defined as a toxic effect in the subject at any dose, cannot be reasonably attributed to the subject's underlying disease, other conditions, and/or concomitants, that the investigator determines to be related (including definitely, likely, or possibly) to the XS005 injection.
Incidence of Adverse Events (AEs) | 4 months
  AE is defined as any adverse medical event within 4 months after the the first infusion of XS005.
Maximum tolerated dose (MTD) | within 7 days after the the first infusion of XS005.
  MTD is defined as the highest dose level of less than or equal to 2 DLT among the 6 subjects finally determined.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From the start of treatment until the time of first disease progression or death , assessed up to 12 months post-treatment
  PFS : defined as the time from the start of treatment until the onset of tumor progression or death from any cause;

CONTACTS AND LOCATIONS:
Locations (1):
- Dushu Lake Hospital Affiliated to Soochow University, Suzhou, Jiangsu, China